CLINICAL TRIAL: NCT01734460
Title: Maternal Sleep Disordered Breathing and Fetal Growth
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: TASMC-12-RT-0510-12-TLV-CTIL
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-08

CONDITIONS: Sleep Disordered Breathing
Keywords: pregnancy, snoring, fetal growth
MeSH Terms: conditions — Sleep Apnea Syndromes; Snoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- third trimester pregnant women: no intervention

SUMMARY:
Sleep disordered breathing (SDB) is a common condition affecting up to 9% of adults with serious neurocognitive, metabolic and cardiovascular consequences that has a significant impact on public health. Evidence indicates that the physiologic changes occurring during pregnancy, particularly during the third trimester, increase the risk of those women to develop SDB. As in the general population, SDB during pregnancy is more frequent among obese women. In the light of the increasing prevalence of obesity among females of reproductive age, SDB may thus have an increasingly significant impact on women's and children's health by contributing to the adverse maternal and fetal outcomes associated with maternal obesity.

Only a limited amount of data is available on the consequences of maternal SDB during pregnancy. Even less information is available on the effect of maternal SDB on fetal growth and development. The current proposal is designed to specifically explore the effect of maternal SDB on fetal growth.

It has been suggested that fetal growth as reflected in birth weight is a strong correlate for conditions occurring in the intrauterine environment with potential long lasting influence on a child's health.

Our overall hypothesis is that the intermittent hypoxia, sleep fragmentation and the metabolic alterations associated with maternal SDB will affect fetal growth.

Using a variety of methods and a multidisciplinary approach, we will explore the following objectives: 1) The effect of maternal SDB on fetal growth ; 2) To explore mechanisms that may underlay the effect of maternal SDB on fetal growth 3) To explore the long term (first 3 years of life) effect of maternal SDB on a child's growth.

The results of this study will make an important contribution to the fields of women and children's health. It will provide better insight into the mechanisms by which disrupted maternal sleep affects fetal growth.

We expect that the findings from our study will enable the defining of a new treatable clinical entity or syndrome: "the infant of the gestational SDB mother", for which early diagnosis and intervention might be of major importance to the newborn infant.

ELIGIBILITY:
Inclusion Criteria:

* low risk third trimester pregnant women

Exclusion Criteria:

* pregnancy complications (preeclampsia, HTN, GDM),
* any chronic medical condition.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: women health care centers
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
birth weight | at birth

SECONDARY OUTCOMES:
birth length | at birth

OTHER OUTCOMES:
birth head circumference | at birth

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel